CLINICAL TRIAL: NCT06511791
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Exploratory Trial to Investigate the Effect of FE 999302 When Administered During Different Time Intervals in Women Undergoing Controlled Ovarian Stimulation With a Fixed Dose of Follitropin Delta in a Gonadotropin-releasing Hormone Antagonist Protocol.
Brief Title: An Exploratory Study to Investigate the Effect of FE 999302 When Given Together With Follitropin Delta at Different Time Intervals During Controlled Ovarian Stimulation.
Acronym: Celestial-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This is a company decision made not related to safety concerns. Rather, it reflects a broader portfolio assessment and the desire to focus on programs that can bring timely and meaningful benefit to patients.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000427; 2023-508149-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin delta

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo Group (Placebo Comparator): Placebo from day 1 to end of stimulation
  Interventions: Drug: Follitropin delta; Drug: Placebo FE 999302
- FE 999302 Group (Active Comparator): FE 999302 from stimulation day 1 to end-of-stimulation
  Interventions: Drug: FE 999302; Drug: Follitropin delta
- FE 999302 and Placebo Group (Active Comparator): FE 999302 from stimulation day 1 to stimulation day 5, and placebo stimulation day 6 to end-of-stimulation
  Interventions: Drug: FE 999302; Drug: Follitropin delta; Drug: Placebo FE 999302
- Placebo and FE 999302 (Active Comparator): Placebo from stimulation day 1 to stimulation 5, FE 999302 from stimulation day 6 to end-of-stimulation.
  Interventions: Drug: FE 999302; Drug: Follitropin delta; Drug: Placebo FE 999302

INTERVENTIONS:
Drug: FE 999302 — Effect on parameters influencing pregnancy rates when administered during different time intervals in women undergoing controlled ovarian stimulation with a fixed dose of follitropin delta in a gonadotropin-releasing hormone (GnRH) antagonist protocol
  Arms: FE 999302 Group; FE 999302 and Placebo Group; Placebo and FE 999302
Drug: Follitropin delta — The effect on parameters influencing pregnancy rates in women undergoing controlled ovarian stimulation with a fixed dose of follitropin.
  Other Names: REKOVELLE
Drug: Placebo FE 999302 — No active ingredient, subcutaneous injection.
  Arms: FE 999302 and Placebo Group; Placebo Group; Placebo and FE 999302

SUMMARY:
This is a phase 1b clinical trial with Choriogonadotropin beta (FE999302) and Follitropin delta (Rekovelle). The trial is a randomised, double blind, placebo controlled, parallel group, exploratory trial, investigating the effect of FE 999302 when administered during different time intervals in women undergoing controlled ovarian stimulation with a fixed dose of follitropin delta in a antagonist protocol.

DETAILED DESCRIPTION:
The trial is multicentre, randomized, partially double-blind, placebo-controlled, parallel-group investigating the effect of FE999302 on parameters influencing pregnancy rates in women undergoing controlled ovarian stimulation with a fixed dose of follitropin.

The primary endpoint is the number of good-quality blastocysts on day 5 after oocyte retrieval. Secondary endpoints are number of follicles by size category and serum concentration of different hormones on stimulation day 6 and end-of stimulation, the number of stimulation days and oocytes retrieved, the number of metaphase II oocytes and fertilised oocytes, number of blastocysts on day 5, number of cryopreserved blastocysts, endometrial thickness at eos, positive bhcg rate, clinical pregnancy, vital pregnancy and ongoing pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject informed consent form signed before any trial-related activities.
2. In good physical and mental health as judged by the investigator.
3. Serum anti-Müllerian hormone (AMH) levels of >35.0 pmol/L at screening (measured at central laboratory).
4. Pre-menopausal women between the ages of 18 and 40 years. The subjects must be at least 18 years (including the 18th birthday) and no more than 40 years (up to the day before the 41st birthday) when they sign the informed consent(s).
5. Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II or with partners diagnosed with male factor infertility, eligible for in vitro fertilisation (IVF) and/or intracytoplasmic sperm injection (ICSI) using fresh or frozen ejaculated sperm from male partner or sperm donor.
6. Infertility for at least 1 year before screening for subjects <35 years or for at least 6 months for subjects ≥35 years (not applicable in case of tubal or severe male factor infertility).
7. No more than two controlled ovarian stimulation cycles initiated, regardless of outcome (taking exclusion criteria 2 and 3 into account) and the subject must be suitable for treatment with 10 or 15 µg/day follitropin delta (corresponding to 150 or 225 IU).
8. Regular menstrual cycles of 24-35 days (both inclusive), presumed to be ovulatory.
9. Early follicular phase (cycle day 2-5) serum levels of follicle-stimulating hormone (FSH) between 1 and 15 IU/L (measured at central laboratory).
10. Body mass index (BMI) between 18.0 and 32.0 kg/m2 (both inclusive) at screening.

Exclusion Criteria:

1. Known polycystic ovary syndrome (PCOS) or known endometriosis stage III-IV (American Society for Reproductive Medicine, 2012).
2. Poor response in a previous controlled ovarian stimulation cycle using a gonadotropin starting dose of 150 IU/day (corresponding to 10 µg follitropin delta) or higher. Poor response is defined as <4 oocytes retrieved, or cycle cancellation before oocyte retrieval due to inadequate follicular development.
3. Severe ovarian hyperstimulation syndrome (OHSS; grade 4 or 5) in a previous controlled ovarian stimulation cycle, as judged by the investigator.
4. One or more follicles ≥10 mm (including cysts) observed on the transvaginal ultrasound before randomisation on stimulation day 1 (puncture of cysts is allowed before randomisation).
5. Any known clinically significant systemic disease (e.g. insulin-dependent diabetes).
6. Any known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver, or kidney) with the exception of controlled thyroid function disease.
7. Known tumours of the ovary, breast, uterus, adrenal gland, pituitary, or hypothalamus which would contraindicate the use of gonadotropins.
8. Any abnormal finding of clinical chemistry and haematology at screening or vital signs at randomisation, which is judged clinically relevant by the investigator and/or requires intervention.
9. Currently breast-feeding.
10. Undiagnosed vaginal bleeding.
11. Findings at the gynaecological examination at screening which preclude gonadotropin stimulation or are associated with a reduced chance of pregnancy, e.g. congenital uterine abnormalities or retained intrauterine device.
12. Pregnancy (negative urinary pregnancy tests must be documented at screening and before randomisation) or contraindication to pregnancy.
13. Use of fertility modifiers during the last menstrual cycle before screening, including dehydroepiandrosterone (DHEA) and metformin or cycle programming with oral contraceptives, progestogen, or estrogen preparations.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Number of good-quality blastocysts | Day 5
  Number of good-quality blastocysts on day 5 after oocyte retrieval

SECONDARY OUTCOMES:
Number and Size of Follicles | Day 5 and up to 20 days
  Number of follicles by size category on stimulation day 5 and at end-of-stimulation
Serum hormone concentrations | Day 5, up to 20 days, and up to 22 days
  Serum hormone concentrations of progesterone, androstenedione, estradiol, inhibin B, and luteinising hormone (LH).
Number of Stimulation Days | Up to 20 days
  Number of stimulation days
Number of Oocytes | Up to 22 days
  Number of oocytes retrieved
Number of metaphase II oocytes | Up to 22 days
  Number of metaphase II (MII) oocytes
Number of fertilised oocytes | Up to 22 days
  Number of fertilised (2 pronuclei [2PN]) oocytes
Number of blastocysts | Up to 27 days
  Number of blastocysts
Number of cryopreserved blastocysts | Up to 28 days
  Number of cryopreserved blastocysts
Endometrial thickness | Up to 20 days and up to 27 days
  Endometrial thickness
Positive βhCG | 13-15 days after fresh transfer
  Positive βhCG
Clinical pregnancy | 5-6 weeks after fresh transfer
  Clinical pregnancy measured by at least one gestational sac 5-6 weeks after fresh transfer
Vital pregnancy | 5-6 weeks after fresh transfer
  Vital pregnancy measured by at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after fresh transfer
Ongoing pregnancy | 10-11 weeks after fresh transfer
  Ongoing pregnancy measured by at least one intrauterine viable fetus 10-11 weeks after fresh transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ferring Pharmaceuticals, Study Director — Ferring Pharmaceuticals
Locations (12):
- Belgium (2):
  - Ferring Investigational Site, Brussels
  - Ferring Investigational Site, Edegem
- Ferring Investigational Site, Prague, Czechia
- Denmark (2):
  - Ferring Investigational Site, Copenhagen
  - Ferring Investigational Site, Hvidovre
- Norway (3):
  - Ferring Investigational Site, Bergen
  - Ferring Investigational Site, Porsgrunn
  - Ferring Investigational Site, Trondheim
- Spain (4):
  - Ferring Investigational Site, Barcelona
  - Ferring Investigational Site, Madrid
  - Ferring Investigational Site, Seville
  - Ferring Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: No